CLINICAL TRIAL: NCT05026138
Title: Natural History, Epidemiology and Pathogenesis of Severe HPV-Related Diseases (Neptune)
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 210029; 21-I-0029
Record Dates: First submitted 2021-08-27; First posted 2021-08-30 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11-24

CONDITIONS: Human Papillomavirus
Keywords: Mucosal Disease; Immunocompromised; Genetic Defects; Infection; Neoplasia; Natural History
MeSH Terms: conditions — Infections; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Biological relatives without HPV: Biological relatives, household contacts, and/or sexual partners without current HPV disease serving as controls to be compared with those from affected participants for evaluation of the differences between people with HPV and without.
- Participants with HPV: Patients with recurrent HPV related diseases refractory to standard-of-care medical or surgical interventions.

SUMMARY:
Background:

Most symptoms of human papillomaviruses (HPV) infection, do not cause serious health problems, but some do. As HPV can cause uncontrolled growth of infected cells, some people can develop benign skin lesions, larger warts, genital lesions, tumors or cysts that do not respond to treatment. Researchers want to learn why.

Objective:

To better understand why some people are more likely than others to get sick from HPV infection, and why medicine or surgery is not always effective.

Eligibility:

People aged 3 years and older who have had multiple outbreaks of HPV-related warts and/or lesions that do not respond to treatment. Healthy relatives are also needed.

Design:

Participants will be screened with a medical history, physical exam, and blood tests.

Participants may have study visits as an outpatient or an inpatient (admitted overnight to the NIH hospital) and be followed over several years by our doctors and researchers at the NIH.

Participants may have a cervical and/or anal Pap test. They may give samples of semen, cervicovaginal secretions, urine, saliva, or stool. Small pieces of skin, the inside of the cheek, and/or the gums may be collected with a punch or scrape biopsy to understand how HPV affect the growth of cells.

Mucus and skin may be collected by rubbing the area with a cotton swab. Collection areas may include the inside the mouth, nostrils, skin, genitals, and/or in or around the anus.

Biopsies may be collected. If participants need to have a biopsy as part of medical care, then we may ask if extra samples can be collected for research. Biopsies we may collect are bone marrow, lymph node, genitals, or in or around the anus.

Participants may have leukapheresis. Blood is taken from a needle placed in one arm. A machine separates out the white blood cells. The rest of the blood is returned through a needle in their other arm.

Samples may be used for genetic tests and/or to make special cells called induced pluripotent stem cells.

Participants may have follow-up visits once a year for 10 years.

Benefits:

We are not testing new HPV treatments in this study and you might not benefit from participating. However, we may learn new information about your condition that we will share with you and your doctor. We may make recommendations for your medical care based on current accepted treatment.

What we learn from you and other participants in this study might help other people. We hope we can use this information to develop new treatments and therapies in the future....

DETAILED DESCRIPTION:
Study Design: This is a prospective, longitudinal natural history study. Total length of individual participation is 10 years.

Primary Objective: To define the clinical, immunologic, and genetic bases of severe disseminated, recurrent, and treatment-refractory HPV-related skin and mucosal disease.

Secondary Objectives:

1. Identify novel genetic defects associated with severe HPV-related diseases.
2. Define the natural history of HPV infections on skin and mucosal tissue in immunocompromised hosts.
3. Define the epidemiology of skin and mucosal HPV variants in immunocompromised hosts by next-generation sequencing.
4. Define the distribution of immune cells in skin and mucosal surfaces of patients with severe HPV-related diseases and

immunologic correlates of HPV-disease progression.

Primary Endpoint: Identify novel immunologic and/or genetic determinants of the susceptibility to severe disseminated, recurrent, and

treatment-refractory HPV-related diseases.

Secondary Endpoints: 1. Identify virologic, clinical, and immunologic predictors of progressive HPV-related diseases.

2. Define the cellular and functional components involved in control or lack thereof of HPV infection in different cutaneous and

mucosal surfaces.

The purpose of this study is to identify clinical and immunologic correlates of increased susceptibility to human papillomavirus (HPV) infections, HPV related dysplasia/cancer, or any other HPV-related clinical manifestations. We will enroll patients with disseminated, multifocal or recurrent HPV-related diseases refractory to standard-of-care medical or surgical interventions. Healthy family members household contacts, and/or sexual partners will also be enrolled as comparators. This protocol will allow long-term follow-up of patients with primary or acquired immunologic abnormalities associated with such increased susceptibility to HPV-related diseases. It will also allow periodic clinical and laboratory evaluation with collection of blood, biological fluids, tissue and mucosal swabs, and tissue biopsies for medically indicated purposes. Additional research studies on these samples will be aimed to identify genetic and immunologic bases of their HPV-related diseases and inform the development of specific and effective treatment interventions.

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion Criteria for All Participants

1. Aged >=3 years (except for household contacts and sexual partners of participants with HPV-related diseases, who must be aged 18 years and older).
2. Able to provide informed consent or, if younger than 18, be accompanied by a parent(s)/legal guardian(s) who is able to provide informed consent.
3. Willing to allow genetic testing on their collected biological samples.

Additional Inclusion Criteria for Participants with HPV-related Diseases

Has severe, disseminated, recurrent, and treatment-refractory HPV infection, defined as one or more of the following confirmed by medical record review or participant health history:

1. In participants without known primary or acquired immunodeficiency:

   1. Multiple skin warts (>=5) recurrent* or refractory to standard-of-care interventions (eg, topical imiquimod, acetylsalicylic acid, cryotherapy, cantharidin, podophyllotoxin, bleomycin, cauterization, cidofovir, fluorouracil).
   2. Concomitant skin warts (irrespective to recurrence or treatment response) AND any historical or current clinical and/or histologic or cytologic evidence of mucosal HPV-related diseases (oral, nasal, laryngeal, vaginal, anal, penile, or cervical).
   3. Mucosal condyloma or other HPV-related diseases that are recurrent* or refractory to standard-of-care interventions.
   4. Historical evidence of mucosal condyloma or any HPV-related diseases occurring irrespective of response to standard-of-care interventions and involving more than one mucosal site.
2. In participants with known primary or acquired immunological defect (including idiopathic CD4 lymphopenia, immunosuppressive treatment, or HIV/AIDS):

   a. Any skin OR mucosal HPV-related diseases
3. In any participant:

   1. Recurrent invasive skin or mucosal HPV-related squamous cell carcinoma (HPV-SCC).
   2. Historical or current histologic evidence of invasive HPV-SCC of any mucosal site in subjects with family history of HPV-SCC in 1 or more family members.

      * The lack of complete response to 2 or more interventions is defined as treatment-refractory disease in the protocol, while the reappearance of a skin or mucosal lesion after complete resolution is defined as recurrence.

Additional Inclusion Criteria for Controls

1. Biological relative, household contact, or sexual partner of the index participant (with HPV-related diseases) who meets one of the following criteria:

1. does not have any historical or current clinical and/or histologic or cytologic evidence of skin or mucosal HPV-related diseases, or
2. has historical or current clinical and/or histologic or cytologic evidence of skin or mucosal HPV-related diseases but does not meet the criteria to be enrolled in this study as a participant with HPV-related disease.

EXCLUSION CRITERIA:

Individuals meeting any of the following criteria will be excluded from study participation:

1. Laboratory abnormalities contraindicating research evaluations and procedures in patients without previous history of cytopenias: neutropenia (absolute neutrophil count <500 cells/microL) or thrombocytopenia (platelets <10,000/microL). Medical record review may be used to for determining eligibility if the laboratory tests were collected <= 90 days prior to the screening visit.
2. Inability to reliably keep research appointments and/or adhere to research procedures.
3. Any condition that, in the opinion of the investigator, contraindicates participation in this study.

Additional Exclusion Criteria for Controls

1. Has HPV-related disease that may indicate enrollment as an affected participant rather than as a healthy biological relative, household contact, or sexual partner.

Co-enrollment guidelines: Participants may be co-enrolled in other studies; however, study staff should be notified of co-enrollment.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants will have HPV infection with severe, disseminated, recurrent, and treatment-refractory HPV related skin and mucosal disease. Healthy biological relatives, household contacts, and/or sexual partners will also be recruited to serve as controls for research tests.
Sampling Method: Probability Sample
Enrollment: 850 (Estimated)
Dates: Start 2021-11-17 (Actual); Primary Completion 2047-03-31 (Estimated); Study Completion 2047-03-31 (Estimated)

PRIMARY OUTCOMES:
Identify novel immunologic and/or genetic determinants of the susceptibility to severe disseminated, recurrent, and treatment-refractory HPV-related diseases. | Throughout the study
  To define the clinical, immunologic, and genetic bases of severe disseminated, recurrent, and treatment-refractory HPV-related skin and mucosal disease.

SECONDARY OUTCOMES:
Identify virologic, clinical, and immunologic predictors of progressive HPV-related diseases | Throughout the study
  Identify novel genetic defects associated with severe HPV related diseases.
Define the cellular and functional components involved in control or lack thereof of HPV infection in different cutaneous and mucosal surfaces | Throughout the study
  Define the natural history of HPV infections on skin and mucosal tissue in immunocompromised hosts; Define the epidemiology of skin and mucosal HPV variants in immunocompromised hosts by next-generation sequencing; Define the distribution of immune cells in skin and mucosal surfaces of patients with severe HPV-related diseases and immunologic correlates of HPV-disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Lisco, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2021-I-0029.html